CLINICAL TRIAL: NCT02273193
Title: Utility Of Hemoglobin A1C (HbA1C) For The Diagnosis Of Gestational Diabetes Mellitus (GDM).
Brief Title: Utility Of Hemoglobin A1C For The Diagnosis Of Gestational Diabetes
Acronym: A1cGDM
Status: Completed | Type: Observational
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FWH20130041H
Record Dates: First submitted 2014-10-14; First posted 2014-10-23 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant Women: Pregnant Women in the first trimester (<13 weeks) of pregnancy and the second trimester of pregnancy.

SUMMARY:
A prospective cohort research study is being conducted in the Mike O'Callaghan Federal Medical Center (MOFMC), Department of Family Medicine, Obstetrics Clinic to determine if early screening with hemoglobin A1C, a blood test for blood glucose, can be used to identify women with hyperglycemia or Gestational Diabetes Mellitus (GDM) in the first semester of pregnancy in place of a fasting blood glucose blood test. This study will also determine how hemoglobin A1C compares with the oral glucose tolerance test (GTT) done as a standard of care with the standard of care second trimester prenatal care testing. Subjects recruited and consented during the Obstetrics Orientation Class will have two (2) additional blood tests drawn with their standard of care prenatal tests in the first trimester (<13 weeks) of pregnancy and at the second trimester (24-28 weeks) of pregnancy. Subjects identified as having GDM by blood HbA1C, fasting glucose or the 2 hr OGTT will be treated for GDM with standard of care by their primary care provider. The correlation of blood HbA1C with the fasting glucose in the first trimester of pregnancy and with the 2 hr OGTT will be determined for early detection and diagnosis of GDM. This study will contribute to understanding the role of HbA1C in pregnancy and the development of GDM.

DETAILED DESCRIPTION:
This is a prospective cohort research study conducted in the Mike O'Callaghan Federal Medical Center (MOFMC), Department of Family Medicine Residency and Obstetrics Clinics. Subjects will be pregnant female active duty or DoD beneficiaries 18 years or older recruited from the MOFMC, Department of Family Medicine Residency Clinic, and Obstetrics Orientation Class at Nellis AFB. At the screening, the Research Assistant discusses the study, answers all questions, obtains Informed Consent, and schedules appointments for routine OB care. The research design includes a screening visit to obtain written consent and two (2) additional laboratory blood tests obtained during the standard of care prenatal screen testing during the first and second trimesters of pregnancy. Each laboratory blood test will be done via 1 venipuncture for 5-10 ml (1-2 teaspoons) of blood. The OB nurse orders all labs upon completion of the Obstetrics Orientation Class.

Screening Visit: Initial Standard of Care Obstetrics Appointment

* Obtain subject signed Informed Consent document and HIPAA Authorization
* Demographic data: age, race, weight, height, estimated week of gestation
* Review past medical history

First Trimester Prenatal Visit (<13 weeks) Screen Testing

* Subjects will have routine prenatal labs drawn to include the HbA1C blood test which is standard of care
* Subjects will have fasting (10 hour) glucose blood test will be ordered along with these labs (research driven)

Second Trimester Prenatal Visit (24-28 weeks)

* Subjects will have routine prenatal labs drawn to include the 2 hr glucose tolerance test (2 hr OGTT) which is standard of care
* Subjects will have will be the HbA1C blood test ordered along with these labs (research driven)

Delivery and Neonatal Data Collection

-Select data regarding delivery and neonatal health will be tracked. All of this data is already routinely collected as standard of care and will be found in the patient record. This will require no interaction with the patient or the neonate

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion:

* Active duty or DoD beneficiaries of childbearing age 18 years or older with a positive pregnancy test (beta human chorionic gonadotropin).

Exclusion:

* Active duty or DoD beneficiaries of childbearing age 18 years or older with a positive pregnancy test (beta human chorionic gonadotropin) known to have and/or develop during the study any of the following upon review of their medical record:

  * Hemoglobinopathy (including sickle cell disease or trait, thalassemia)
  * Chronic kidney disease
  * Diabetes
* Active duty or DoD beneficiaries of childbearing age 18 years or older with a positive pregnancy test (beta human chorionic gonadotropin) taking any of the following:
* Erythropoietin
* Daily oral steroids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active duty or DoD beneficiaries of childbearing age 18 years or older with a positive pregnancy test
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Fasting Glucose will be obtained during the first trimester of pregnancy | 13 weeks

SECONDARY OUTCOMES:
Hemoglobin A1c will be obtained during the second trimester of pregnancy (between 24-28 weeks) | 24-28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crawford, MD, Principal Investigator — Mike O'Callaghan Federal Medical Center
Locations (1):
- Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No